CLINICAL TRIAL: NCT03358563
Title: Pilot Neoadjuvant Trial of Chemohormonal Therapy Followed by Prostatectomy in Patients With High Risk or Oligometastatic Prostate Cancer
Brief Title: Pilot Trial of Chemohormonal Therapy Followed by Prostatectomy in High Risk Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW17009; 2017-0606 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2017-02428 (Registry Identifier: NCI Trial ID); Protocol Version 1/18/2022 (Other: UW Madison)
Record Dates: First submitted 2017-10-13; First posted 2017-11-30 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatectomy; Chemohormonal therapy; Androgen deprivation therapy; docetaxel chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Degarelix SC + bicalutamide + docetaxel (Experimental): Degarelix SC monthly x3 + bicalutamide 50mg orally QD x 14 wks + Docetaxel 75mg/m2 IV q 21 days x 3
  Interventions: Drug: Docetaxel; Drug: Degarelix; Drug: Bicalutamide
- DegarelixSC + bicalutamide + docetaxel + Ferumoxytol enhanced MRI (Experimental): Degarelix SC monthly x3 + bicalutamide 50mg orally QD x 14 wks + Docetaxel 75mg/m2 IV q 21 days x 3 + Ferumoxytol enhanced MRI within 21 days prior to start of hormonal therapy and second and final ferumoxytol-enhanced MRI at the conclusion of hormone therapy but prior to their prostatectomy.
  Interventions: Drug: Docetaxel; Drug: Degarelix; Drug: Bicalutamide; Radiation: Ferumoxytol-enhanced MRI imaging

INTERVENTIONS:
Drug: Docetaxel — Docetaxel is a commercially marketed product that has been approved by the FDA for the treatment of metastatic prostate cancer. It is also approved for the treatment of other malignant disease, such as locally advanced or metastatic breast cancer that returns after any prior chemotherapy; locally advanced or metastatic non-small cell lung cancer that recurs after prior platinum-based chemotherapy. However, the FDA does not currently approve its use in patients with localized prostate cancer but no evidence of radiographic metastases.
  Other Names: docetaxel chemotherapy; taxotere; PR 56976; NSC #628503
Drug: Degarelix — Degarelix is a leuteinizing hormone-releasing hormone (LHRH) antagonist. Degarelix is administered at an initial dose of 240 mg subcutaneously (2 separate injections of 120mg each totaling 240 mg) two weeks prior to cycle 1 day 's 1 treatment with chemotherapy. The initial dose is followed by a maintenance dose of 80mg administered subcutaneously as a single injection every 28 days at cycle 2 day 1 (+/- 7 days) and cycle 3 day 10 (+/- 7 days)
  Other Names: Degarelix acetate
Drug: Bicalutamide — The dose for bicalutamide tablets therapy in combination with an LHRH analog is one 50 mg tablet once daily (morning or evening), with or without food. It is recommended that bicalutamide tablets be taken at the same time each day. Treatment with bicalutamide tablets should be started at the same time as treatment with an LHRH analog.
  Other Names: Casodex
Radiation: Ferumoxytol-enhanced MRI imaging — Ferumoxytol-enhanced MRI imaging will evaluate immune micro-environment in the prostate. Three subjects enrolled to the study will undergo the first ferumoxytol-enhanced MRI imaging within 21 days prior to start of hormonal therapy followed by second and final ferumoxytol-enhanced MRI at the conclusion of hormone therapy but prior to their prostatectomy.
  Arms: DegarelixSC + bicalutamide + docetaxel + Ferumoxytol enhanced MRI

SUMMARY:
This is a pilot multimodality treatment approach trial with androgen deprivation therapy in combination with docetaxel chemotherapy followed by radical prostatectomy in patients with newly diagnosed high-risk and oligometastatic prostate cancer. This study aims to evaluate the rates of complete pathologic response (pCR) at the time of prostatectomy as well as PSA response, time to PSA recurrence and safety and toxicity of the combination. This study will be heavily embedded with biomarker analyses of the tumor and tumor cells in circulation as well in the bone marrow before and after treatment and will also include imaging analyses using a novel positron emission tomography (PET) imaging technology.

DETAILED DESCRIPTION:
Per a protocol amendment approved on 9/5/2019 - two ferumoxytol MRI scans were added for 3 participants, represented here as an additional arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without signet cell or small cell features.
* High risk prostate cancer defined as extracapsular extension (cT3a) or seminal vesicle involvement (cT3b) or invasion of adjacent structures (cT4), serum PSA greater than 20 ng/mL or Gleason score of 8 to 10 and/or regional lymph node or
* Oligometastatic disease defined as disseminated metastases beyond regional lymph nodes that meet the following criteria:

  * No visceral metastases
  * Less than four bony metastases.
* Ability to comply with all study procedures and willingness to remain supine for 120 minutes during imaging.
* Patients must be informed of the experimental nature of the study and its potential risks, and must sign an Institutional Review Board (IRB)-approved written informed consent form indicating such an understanding.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
* Patients must be considered candidates for prostatectomy as per standard of care.
* Adequate hematologic and renal function as evidenced by the following within 4 weeks of day 1:

  * ANC greater than or equal to 1500/mm3
  * Hemoglobin (HgB) greater than or equal to 10.0 gr/dL independent of transfusion
  * Platelets greater than or equal to 100,000/mm3
  * Creatinine less than or equal to 2.0 mg/dL
  * Total bilirubin less than or equal to Upper Limit of Normal (ULN)
* Estimated life expectancy of greater than or equal to 12 months at screening.
* Throughout the study, patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) from screening through 3 months after last dose of study drug. Two acceptable methods of birth control thus include the following:

  * A condom (barrier method of contraception) AND One of the following is required:
  * Established and ongoing use of oral, injected, or implanted hormonal method of contraception by the female partner
  * Placement of an intrauterine device or intrauterine system by the female partner
  * Additional barrier method: Contraceptive sponge or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female partner
  * Tubal ligation in the female partner performed at least 6 months before screening
  * Vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy), performed at least 6 months before screening
* While receiving chemotherapy, the patient must use a condom if having sex with a pregnant woman.
* Must agree not to donate sperm from first dose of study drug through 3 months after the last dose of study drug.

Exclusion Criteria:

* Prior treatment for prostate cancer, including ADT, orchiectomy, antiandrogens, ketoconazole, abiraterone acetate or enzalutamide.
* Prior radiation to the prostate.
* Use of other investigational agent for prostate cancer.
* No active secondary malignancy
* Chronic liver disease or abnormal liver function:

  * Total bilirubin greater than ULN (NOTE: in subjects with Gilbert's syndrome, if total bilirubin is greater than ULN, measure direct and indirect bilirubin and if direct bilirubin is within normal range, subject may be eligible) or
  * Alanine (ALT) or aspartate (AST) aminotransferase greater than 2.0 x ULN or
  * ALT or aspartate AST greater than 1.5 x ULN concomitant with alkaline phosphatase greater than 2.5 x ULN.
* Peripheral neuropathy grade greater than 1.
* Active cardiac disease defined as active angina, symptomatic congestive heart failure, or myocardial infarction within the previous 6 months.
* Major surgery within 4 weeks before screening.
* Patients with known psychological or sociological conditions, addictive disorders or family problems, which would preclude compliance with the protocol.
* Herbal supplements that have been shown to modulate testosterone or androgen signaling (e.g. Saw Palmetto) are not allowed while on study.
* Subjects may not be enrolled concurrently on other treatment studies. Any concurrent disease, infection, or comorbid condition that interferes with the ability of the patient to participate in the trial; places the patient at undue risk; or complicates the interpretation of the data, in the opinion of the investigator or medical monitor.
* Subjects who will be receiving Ferumoxytol MRI tracer must:

  * Not have any known hypersensitivity to Feraheme or any of its components
  * Must not have a history of allergic reaction to any intravenous iron product.
  * Must not have a known iron overload (based on medical history)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Change in pCR rates | Up to 6 months
  Evaluate the pathologic complete response (pCR) rates in the primary tumor from patients with newly diagnosed locally advanced or oligometastatic prostate cancer treated with combination androgen deprivation therapy (ADT) and 3 cycles of docetaxel chemotherapy followed by prostatectomy.

SECONDARY OUTCOMES:
Change in PSA | From baseline (3 months prior to prostatectomy) to 4-6 weeks after prostatectomy.
  Evaluate the percentage of change in prostate-specific antigen (PSA) from baseline (3 months prior to prostatectomy) to week 6 after prostatectomy in patients with newly diagnosed locally advanced or oligometastatic prostate cancer treated with combination ADT and docetaxel as well as the maximum decline in PSA that occurs at any point during treatment.
PSA Recurrence | Up to 12 months
  Rate of patients with PSA recurrence at month 12 after surgery
Safety and tolerability of combination ADT and docetaxel measured by CTCAE v.4.0 | Up to 6 months
  Evaluate safety and tolerability of the combination of ADT and docetaxel for up to three months following the last dose of docetaxel.

OTHER OUTCOMES:
Evaluating PSMA PET/MRI imaging | Up to 12 months
  Evaluate PSMA PET/MRI imaging as a method for determining treatment response in primary prostate cancer and metastatic lesions after ADT and docetaxel.
Evaluating Response Heterogeneity | Up to 6 months
  Evaluate heterogeneity of response in multifocal prostate lesions at the time the primary objective is assessed
Change in total tumor burden in individual lesions | Up to 12 months
  Evaluate change in total tumor burden in individual lesions and across all lesions over time for each patient
Evaluating immune microenvironment in prostate with ferumoxytol-enhanced MRI relaxometry | Up to 12 months
  Evaluate immune microenvironment in prostate with ferumoxytol-enhanced MRI relaxometry
Disease progression | Up to 12 months
  Correlate disease progression on MRI, technetium Tc 99m medronate (99mTc-MDP) bone scintigraphy and CT scans with PSMA uptake measures
PSMA PET results and PSA response correlation | Up to 12 months
  Correlate prostate-specific membrane antigen (PSMA) PET results with PSA response and time to PSA progression
Evaluate genomic signatures in multifocal prostate cancer after ADT and Docetaxel | Up to 12 months
  Prostate cancer cells extracted from the prostatectomy specimen will undergo nucleic acid extraction. DNA will be isolated and sequenced using the Foundation Medicine Next Generation Sequencing platform or other genomic panels
Evaluate gene expression signatures in multifocal prostate cancer after ADT and Docetaxel | Up to 12 months
  Prostate cancer cells will be extracted from the prostatectomy specimen and undergo nucleic acid extraction. mRNA will be isolated and analyzed with gene expression panels with quantitative RT PCR and/or next generation sequencing.
Evaluate gene expression signatures in prostate stroma after ADT and Docetaxel | Up to 12 months
  Prostate stromal cells will be extracted from the prostatectomy specimen and undergo nucleic acid extraction. mRNA will be isolated and analyzed with gene expression panels with quantitative RT PCR and/or next generation sequencing.
Evaluate infiltrating immune cells in prostatectomy specimens after ADT and Docetaxel | Up to 12 months
  Immune cells will be extracted from the prostatectomy specimen and bone marry biopsies. These cells are labelled with antibodies and quantified using flow cytometry.
Evaluating EpCAM-positive disseminated and circulating tumor cells | Up to 12 months
  Evaluate epithelial cell adhesion molecule (EpCAM)-positive disseminated and circulating tumor cells for subcellular localization of the androgen receptor and glucocorticoid receptor
Disseminated and circulating tumor cell analyses versus PSMA PET/MRI and clinical outcomes | Up to 12 months
  Correlate disseminated and circulating tumor cell analyses with the PSMA PET/MRI measures and clinical outcomes.
Evaluate immune microenvironment in bone marrow after ADT and Docetaxel | Up to 12 months
  Immune cells will be extracted from the prostatectomy specimen and bone marrow biopsies.
Evaluate secretory profile of stroma after ADT and Docetaxel | Up to 12 months
  Prostate stromal cells will be extracted from the prostatectomy specimen and undergo nucleic acid extraction.
Evaluate immune microenvironment in prostate after ADT and Docetaxel | Up to 12 months
  Evaluating immune microenvironment in prostate by assessing protein and molecular biomarkers after ADT and Docetaxel. Archival formalin-fixed-paraffin-embedded prostate tissue will be used for this aim.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Kyriakopoulos, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Homepage — http://www.uwhealth.org/uw-carbone-cancer-center/47424